CLINICAL TRIAL: NCT06846879
Title: Evaluation of the Quality of Care in the Emergency Department by Studying the Appropriateness of Hospitalizations: Validation of an Algorithm Based on Computerized Hospital Databases
Brief Title: Evaluation of the Quality of Care in the Emergency Department by Studying the Appropriateness of Hospitalizations
Status: Not yet recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: START
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Quality of Care; Evaluation; Emergency Department; Appropriateness
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elegible population: All patients aged 18 years and over who arrived at participating centres between 1 January 2023 and 31 December 2024.

SUMMARY:
The aim of this study is to develop, study and validate a rigorous and sustainable method for assessing the clinical appropriateness of the decision taken in the Emergency Department to admit or not to admit patients.

DETAILED DESCRIPTION:
The information normally recorded in the Emergency Department medical record will be used, as well as the available clinical and administrative databases. For reasons of feasibility, the investigators will also restrict the analysis to patients coming to the Emergency Department with non-specific manifestations in the pulmonary, cardiovascular and abdominal districts, represented by one or more of the following symptoms: dyspnoea, chest pain, transient loss of consciousness, abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

All patients aged 18 years and over who arrived at participating centres between 1 January 2023 and 31 December 2024.

Exclusion Criteria:

All patients under 18 years of age arriving at participating centers between January 1, 2023 and December 31, 2024 and all patients arriving at participating centers outside the time frame January 1, 2023 - December 31, 2024.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 years and over who arrived at participating centres between 1 January 2023 and 31 December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 240000 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Qualitative validation and first refinement of the classification algorithm | From August 2025 to November 2025
  In this first phase of the project, representatives of doctors and nurses from participating hospitals will be asked to express their opinion on content validity. This refers to the accuracy with which a measurement tool covers all aspects of the construct under examination. Its measurement is generally based on the judgment of experts in the field, who are asked to provide feedback on how closely the measurement tool corresponds to the different domains associated with the construct.
  The evaluation will be conducted according to the consensus conference approach, an approach that reduces the risk of excessive subjectivity, intrinsic to content validity. This evaluation will lead to a possible refinement of the individual criteria that make up the algorithm.
Quantitative validation and second refinement of the classification algorithm | From September 2025 to October 2026
  In this second phase, the criterion validity of the algorithm developed in the previous phase will be examined. Criterion validity measures the relationship between the results obtained with the test in question and those obtained with a consolidated reference standard (the criterion, or gold standard) that measures the same construct.
Application of the algorithm to all eligible patients | From November 2026 to Dicember 2026
  Once perfected, the algorithm will be applied to all eligible patients arriving at the ER of participating hospitals within a 24-month period (from January 2023 to December 2024). This means that, for all hospitalized patients, it will be possible to obtain data on the appropriateness of this choice and monitor the evolution of this data over time.
Feasibility of assessing the appropriateness of discharge from the emergency room | From November 2026 to June 2027
  In this phase, an attempt will be made to obtain the data necessary to evaluate the appropriateness of discharges from the ED for eligible patients who were discharged between January 2023 and December 2024. Data will be collected on all accesses in the period considered in order to identify any multiple patient accesses (return visits) and the related presentation tables.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Luigi Gonzaga, Orbassano, Italy

IPD SHARING:
Plan to Share IPD: Undecided